CLINICAL TRIAL: NCT06950398
Title: Normothermic Oxygenated Perfusion (NMP) Viability Testing Before Transplantation of Discarded Livers. An Open Label, Non-randomized, Prospective, Single Arm Trial
Brief Title: Normothermic Oxygenated Perfusion (NMP) Viability Testing Before Transplantation of Discarded Livers
Acronym: TRANSPERF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 35RC22_9768_TRANSPERF
Record Dates: First submitted 2024-11-19; First posted 2025-04-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Organ Transplantation; Liver Dysfunction; Liver Diseases
Keywords: Liver Transplantation; Normothermic oxygenated perfusion; NMP; Discarded livers; Viability assessment
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: National, multicenter, exploratory open-label, prospective, non-randomized, single-arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normothermic oxygenated perfusion (NMP) viability testing (Experimental): Discarded liver grafts are connected to a normothermic perfusion machine (OrganOx Metra®) for a period of 4 to 12 hours prior to transplantation, to assess their viability.
  Interventions: Other: NMP viability testing

INTERVENTIONS:
Other: NMP viability testing — NMP viability testing before transplantation of discarded livers

SUMMARY:
Liver transplantation (LT) is a highly effective treatment for end-stage liver disease and early-stage primary liver cancer. As such, the demand for donor livers greatly exceeds supply; in 2021 in France, 12.9% of patients on the waitlist either died or were delisted for worsening of their condition.

However a substantial number of perfectly viable organs are wrongly discarded based on a highly subjective assessment as the level of acceptance varies widely depending on the physician's judgement.

The idea of using Normothermic Machine Perfusion (NMP) not only to preserve the liver graft but also for selection purposes is a concept that has been already investigated. A few trials have analyzed the value of normothermic perfusion to assess rejected liver grafts.

Several teams demonstrated that NMP provides a tool to assess organ viability pre-transplantation as the liver is able to maintain an almost physiological metabolism.

These preliminary results came from small samples, 45% of which originated from donation after circulatory death (DCD). They need confirmation in a larger sample of organs from donors with brainstem death (DBD), adapted to the French liver allocation system.

This trial will reproduce and confirm the results of the previous studies in order to establish viability testing as the de facto method for high-risk or rejected grafts. It will also validate existing viability markers so as to define a new standard for viability testing using NMP.

DETAILED DESCRIPTION:
Liver transplantation (LT) is a highly effective treatment for end-stage liver disease and early-stage primary liver cancer. As such, the demand for donor livers greatly exceeds supply; in 2021 in France, 12.9% of patients on the waitlist either died or were delisted for worsening of their condition.

Demand for liver grafts has driven the wider use of extended criteria donors (ECD). Grafts from ECD donors are associated with an increased risk of primary non-function, which is difficult to predict on an individual basis. The suitability of donor livers is determined based on donor history, age, weight, biological parameters of liver function, radiologic features, as well as the graft's macroscopic aspect at the time of procurement. The predictive value of these parameters to detect grafts unsuitable for transplantation is low, especially in the group of grafts obtained from ECD. Hence, the viability of donor livers can only be assessed after the fact, which could be life threatening for recipients of ECD livers.

As a result, a substantial number of perfectly viable organs are wrongly discarded based on a highly subjective assessment as the level of acceptance varies widely depending on the physician's judgement. In France, 253 (20%) of proposed livers were rejected in 2021.

Per current practices, livers are made available for rescue allocation after 5 refusals from 5 different transplant centers before being definitely discarded. Although the reasons for refusal are sometimes evident, (i.e. suspicious tumor or cirrhosis on the donor's CT-scan), most of the time refusal is based on the donor's clinical and biological characteristics.

This multicentric prospective non-randomized trial aims to evaluate the potential of NMP to provide an objective viability assessment of discarded livers. The co-primary endpoints will be (i) the rate of initially discarded livers eventually rescued after evaluation on a normothermic machine and (ii) the rate of functional grafts at 3 months among transplanted rescued livers.

A graft is considered functional at 3 months if the recipient remains alive and no retransplantation has been necessary within that period.

The device that will be used to perfuse the grafts is the OrganOx metra. It perfuses the donor liver with blood, oxygen and nutrients, as well as a number of medications (bile salt, insulin, heparin and prostacyclin), at normal body temperature to mimic ideal physiological conditions and preserve the organ for up to 24 hours. The device provides information as to the haemodynamic, synthetic and metabolic function of the liver to assist the clinician in assessing the organ's suitability for transplantation.

For a liver to be considered viable it has to meet specific viability criteria that are easily assessed using the perfusion device. Several teams demonstrated that NMP provides a tool to assess organ viability pre-transplantation as the liver is able to maintain an almost physiological metabolism. This is especially important as NMP allows an objective assessment of grafts driving the decision to transplant based upon actual graft function rather than a rather superficial risk assessment, which is what is being done currently. Mergental et al. proposed in 2016 lactate clearance (i.e. < 2.5 mmol/l) as a marker of viability in high-risk or discarded livers while Watson et al. suggested that viability is a combination of several characteristics including transaminases, glucose metabolism, lactate clearance, and acid-base balance. In addition, the ability of the liver to maintain acid-base homeostasis was shown to be predictive of post-operative outcomes. Sutton et al. also suggested that bile output may differentiate viable from non-viable livers. Other proposed criteria include hemodynamic parameters (hepatic artery and portal vein flow) and bile composition during NMP.

In 2020, Mergental et al. reported validation of lactate clearance as a viability criteria (i.e. < 2.5 mmol/l within 4 hours) allowing transplantation to be performed using 22 of 31 discarded livers with 100% 90-day survival. Another trial reported successful transplantation after NMP using a custom-built device of 15 livers out of 21 discarded grafts. These preliminary results came from small samples, 45% of which originated from donation after circulatory death (DCD). They need confirmation in a larger sample of organs from donors with brainstem death (DBD), adapted to the French liver allocation system. Grafts from DCD donors will not be included because, in France, DCD donors are subjected to in situ normothermic regional perfusion before procurement. Only liver grafts procured from DBD donors will be included in this study.

ELIGIBILITY:
INCLUSION CRITERIA :

FOR LIVER DONORS

* Donation after brainstem death (DBD)
* Liver graft refused by 5 different transplant centres and after rescue allocation ("hors tour")

FOR LIVER TRANSPLANT RECIPIENTS

* ≥ 18 years old
* Candidates for a first elective liver transplantation (patients with a pre-transplant work-up excluding: re-transplantation, emergency transplantation (e.g. fulminant hepatitis), multi-organ or heterotopic transplantation)
* UNOS status IV (non-ventilated, no vasopressor support)
* Absence of renal insufficiency defined as a GFR of less than 60 mL/min/1.73 m² for three months or more
* MELD Score ≤ 25
* Willing and able to attend follow-up examinations
* Having signed an informed consent document

NON-INCLUSION CRITERIA:

FOR LIVER DONORS

* Macroscopic features of advanced fibrosis or cirrhosis at procurement
* Transplantation using a split graft, in situ or ex situ
* Estimated cold ischemic time greater than 8 hours (5 hours maximum of graft transport in cold ischemia)

FOR LIVER TRANSPLANT RECIPIENTS

* Mentally or legally incapacitated
* Transplantation for fulminant hepatic failure
* Early or late re-transplantation
* Combined liver transplant with any other organ, en-bloc or not
* Heterotopic liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
- To assess the efficacy of NMP to provide objective assessment of the viability of livers which were initially discarded | Day 0
  - Rate of initially discarded livers eventually transplanted after viability testing using NMP
  (A stopping rule will be implemented based on the incidence of initially discarded livers eventually transplanted. NMP would be considered as:
  * uninteresting if the rate of discarded livers finally rescued is ≤ 25%
  * and promising if ≥ 40%.)
- To assess grafts survival of rescued livers after transplantation | Month 3, among transplanted rescued livers
  - Rate of functional grafts

SECONDARY OUTCOMES:
- To assess early graft dysfunction | Day 7
  Rate of early allograft dysfunction (EAD). EAD is defined according to Olthoff criteria by the presence of at least one of the following criteria:
  * bilirubin level over 171 mmol/L on PTD7,
  * International Normalized Ratio (INR) over 1.6 on PTD7,
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels > 2000 IU/L within the first 7 PTDs
- To assess primary non-function | Day 7
  Need for re-transplantation and/or death of recipient from liver failure
- To assess intraoperative morbidity | Day 0
  Rate of incidents during reperfusion
- To assess postoperative morbidity | Month 3
  Rate of adverse event and severity, graded according to the Clavien-Dindo classification
- To assess infectious complications | Month 3
  Rate of post-operative pulmonary or surgical site infections
- To assess acute kidney injury | Month 3
  Rate of requirement of renal replacement therapy
- To asses biliary complications | Month12
  Rate of biliary strictures, anastomotic and non-anastomotic, bile duct leaks
- To assess vascular complications | Month 3
  Rate of vascular complications (bleeding, hepatic artery stenosis, hepatic artery thrombosis, portal vein thrombosis, portal vein stenosis)
- To assess acute rejection risks | Month 3
  Rate of biopsy-proven acute rejection
- To assess the need for re-operation | Month 3
  Rate of re-operation (re-laparotomy and/or laparoscopy)
- To assess lengths of stay | Month12
  Median length of intensive care unit stay (days)
- To assess graft survival | Month12
  Time from liver transplantation to re-transplantation or patient death
- To assess recipient survival | Month12
  The time from liver transplantation to death

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - APHP_Hôpital Beaujon, Clichy
  - Hôpital Croix Rousse, Lyon
  - CHU de Montpellier, Montpellier
  - CHU de Rennes PONTCHAILLOU, Rennes
  - CHRU Tours, Tours
  - APHP_Hopital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No